CLINICAL TRIAL: NCT05195099
Title: Effectiveness of a Physiotherapy Respiratory and Neurorehabilitation Treatment Protocol in Patients With COVID-19.
Brief Title: Respiratory Physiotherapy and Neurorehabilitation in Patients With Post-covid19 Sequelae.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal Investigator, Universidad Católica de Ávila
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/01/2022
Record Dates: First submitted 2022-01-14; First posted 2022-01-18 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-01

CONDITIONS: COVID-19 Pandemic
Keywords: coronavirus; physiotherapies techniques; physiotherapies specialty; agnosia for taste; breathing exercises
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator)
  Interventions: Other: respiratory treatment
- respiratory treatment (Experimental)
  Interventions: Other: respiratory treatment

INTERVENTIONS:
Other: respiratory treatment — Respiratory treatment based on aerobic exercise and treatment of the musculature to reduce dyspnoea and increase the capacity for exertion, neurorehabilitative treatment focusing on the sense of smell and taste to on the sense of smell and taste to increase sensitivity in post Covid-19 subjects.

SUMMARY:
The objectives are to reduce dyspnoea, increase exertional capacity, increase vital capacity and respiratory muscle strength.

vital capacity and respiratory muscle strength. In addition to increasing the sensibility of smell and taste, observing if there is a relationship between the decrease of these senses with the senses with appetite and whether appetite has normalised in post-SARS-CoV-2 patients. It is a randomised and blinded experimental study with a control group where the sample recruited will be 30 patients, with a range of of 30 patients, with an age range of 19-42 years, where they carried out an assessment of spirometry, modified Borg dyspnoea scales and modified Medical Research Council (MMRC), Singapure (MMRC), Singapore Smell and Taste Questionnaire (SSTQ) and weekly smell and taste questionnaire.

taste questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* age range between 18 and 42 years.
* patients with respiratory sequelae post Covid-19.
* patients with smell and taste sequelae post Covid-19.

Exclusion Criteria:

* Under 18 years old.
* Over 42 years old.
* Patients not diagnosed with Covid-19 (PCR positive).

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
assessment of spirometry. | 1 year
  modified Borg dyspnoea scales (0, minimum to 10 maximum rated numerical score used to measure dyspnea as reported by the patient during submaximal exercise and is routinely administered during six-minute walk testing)
smell and taste | 1 week
  smell and taste questionnaire, maximum score (maximum capacity) 40 points. 0 minimum

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Ávila, Ávila, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lu Y, Li X, Geng D, Mei N, Wu PY, Huang CC, Jia T, Zhao Y, Wang D, Xiao A, Yin B. Cerebral Micro-Structural Changes in COVID-19 Patients - An MRI-based 3-month Follow-up Study. EClinicalMedicine. 2020 Aug;25:100484. doi: 10.1016/j.eclinm.2020.100484. Epub 2020 Aug 3. PMID 32838240
- [Result] Alawna M, Amro M, Mohamed AA. Aerobic exercises recommendations and specifications for patients with COVID-19: a systematic review. Eur Rev Med Pharmacol Sci. 2020 Dec;24(24):13049-13055. doi: 10.26355/eurrev_202012_24211. PMID 33378057
- [Result] Damm M, Pikart LK, Reimann H, Burkert S, Goktas O, Haxel B, Frey S, Charalampakis I, Beule A, Renner B, Hummel T, Huttenbrink KB. Olfactory training is helpful in postinfectious olfactory loss: a randomized, controlled, multicenter study. Laryngoscope. 2014 Apr;124(4):826-31. doi: 10.1002/lary.24340. Epub 2013 Sep 19. PMID 23929687
- [Result] Altundag A, Cayonu M, Kayabasoglu G, Salihoglu M, Tekeli H, Saglam O, Hummel T. Modified olfactory training in patients with postinfectious olfactory loss. Laryngoscope. 2015 Aug;125(8):1763-6. doi: 10.1002/lary.25245. Epub 2015 Jun 2. PMID 26031472
- [Result] Lechien JR, Chiesa-Estomba CM, De Siati DR, Horoi M, Le Bon SD, Rodriguez A, Dequanter D, Blecic S, El Afia F, Distinguin L, Chekkoury-Idrissi Y, Hans S, Delgado IL, Calvo-Henriquez C, Lavigne P, Falanga C, Barillari MR, Cammaroto G, Khalife M, Leich P, Souchay C, Rossi C, Journe F, Hsieh J, Edjlali M, Carlier R, Ris L, Lovato A, De Filippis C, Coppee F, Fakhry N, Ayad T, Saussez S. Olfactory and gustatory dysfunctions as a clinical presentation of mild-to-moderate forms of the coronavirus disease (COVID-19): a multicenter European study. Eur Arch Otorhinolaryngol. 2020 Aug;277(8):2251-2261. doi: 10.1007/s00405-020-05965-1. Epub 2020 Apr 6. PMID 32253535
- [Result] Wang TJ, Chau B, Lui M, Lam GT, Lin N, Humbert S. Physical Medicine and Rehabilitation and Pulmonary Rehabilitation for COVID-19. Am J Phys Med Rehabil. 2020 Sep;99(9):769-774. doi: 10.1097/PHM.0000000000001505. PMID 32541352
- [Derived] Sanchez Mila Z, Rodriguez Sanz D, Martin Nieto A, Jimenez Lobo A, Ramos Hernandez M, Campon Chekroun A, Frutos Llanes R, Barragan Casas JM, Velazquez Saornil J. Effects of a respiratory and neurological rehabilitation treatment plan in post Covid-19 affected university students. Randomized clinical study. Chron Respir Dis. 2024 Jan-Dec;21:14799731241255967. doi: 10.1177/14799731241255967. PMID 38752418